CLINICAL TRIAL: NCT04374110
Title: Prospective Monitoring of Drug Safety and the Occurrence of Complications During Hospitalization in Patients With Cardiovascular Diseases With COVID-19
Brief Title: Drug Safety and the Occurrence of Complications During Hospitalization in Patients With COVID-19
Acronym: COR-CARDIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 1860/2020
Record Dates: First submitted 2020-04-22; First posted 2020-05-05 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: COVID; Hypertension; Cardiovascular Diseases; Cardiovascular Risk Factor
Keywords: Angiotensin converting enzyme inhibitors; Angiotensin 2 receptor blockers; Renin angiotensin system; COVID-19; Hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hospitalized patients with COVID-19: Hospitalized patients with COVID-19 will be included in the study in centers around Poland.
  Interventions: Other: Clinical data
- Infected SARS-CoV-2 patients: patients with SARS-CoV-2 infection not requiring hospitalization
  Interventions: Other: Clinical data
- Controls: structure-matched and co-existing disease matched control group from the general population.
  Interventions: Other: Clinical data

INTERVENTIONS:
Other: Clinical data — Clinical characteristics from medical records

SUMMARY:
Hospitalized patients with COVID-19 will be included in the study in centers around Poland. After the hospitalization, a short questionnaire will be completed, including pre-hospitalization diagnoses, pre-hospitalization medications, clinical status on admission, the course, complication and the duration of hospitalization. The questionnaire will be available in paper form and on-line.

DETAILED DESCRIPTION:
SARS-Cov-2 infection is characterized by a varied clinical course, from asymptomatic to severe respiratory failure in the course of pneumonia, which can be fatal. There are reports in the literature regarding the relationship between the course of an acute respiratory disease syndrome caused by SARS-CoV-2 virus infection (Coronavirus 2019, COVID-19) and the history of cardiovascular diseases (CVD), including hypertension. It is postulated that the shared element of the pathogenesis of CVD, hypertension and COVID-19 is the renin-angiotensin system and one of its elements, the angiotensin converting enzyme 2 (ACE2). It has been postulated by some authors that in the course of hypertension and antihypertensive treatment with renin-angiotensin system inhibitors, there may be an upregulation of ACE2, which in turn may be related to a higher risk of more severe course of COVID-19. On the other hand there is also data the renin-angiotensin system inhibitors by increasing ACE2 concentration may be protective in the course of severe pneumonia.

The study undertaken by the National Institute of Cardiology aims to assess the safety of the cardiovascular drugs in relation to the occurrence of complications during hospitalization in patients with CVD and COVID-19 infection. The study is being conducted by Polish-German collaboration and was initiated by prof Reinhold Kreutz from Institute of Clinical Pharmacology and Toxicology, Charite, Berlin, Germany and team from National Institute of Cardiology lead by prof. Andrzej Januszewicz and prof. Tomasz Hryniewiecki, Director of the National Institute of Cardiology.

Hospitalized patients with COVID-19 will be included in the study in centers around Poland. After the hospitalization, a short questionnaire will be completed, including pre-hospitalization diagnoses, pre-hospitalization medications, clinical status on admission, the course, complication and the duration of hospitalization. The questionnaire will be available in paper form and on-line.

It will also be planned to include control groups from the official databases: 1) patients with SARS-CoV-2 infection not requiring hospitalization, and 2) structure-matched and co-existing disease matched control group from the general population.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients with COVID-19

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with COVID-19 will be included in the study in centers around Poland.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-06-24 (Estimated); Study Completion 2021-08-24 (Estimated)

PRIMARY OUTCOMES:
Adverse events | through study completion, an average of 2 weeks
  Death, myocardial infarction, heart failure, myocarditis, acute renal failure, stroke

SECONDARY OUTCOMES:
Number of participants with death, myocardial infarction, heart failure, myocarditis, acute renal failure, stroke | through study completion, an average of 2 weeks
  Number of participants with death, myocardial infarction, heart failure, myocarditis, acute renal failure, stroke analyzed separately for each of the endpoints
Ventilation during hospitalization | through study completion, an average of 2 weeks
  Ventilation during hospitalization
Number of participants with death, myocardial infarction, heart failure, myocarditis, acute renal failure, stroke | prolonged follow up, through study completion, an average of one year
  Number of participants with death, myocardial infarction, heart failure, myocarditis, acute renal failure, stroke analyzed separately for each of the endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Januszewicz, MD, PhD, Principal Investigator — National Institute of Cardiology; Tomasz Hryniewiecki, MD, PhD, Principal Investigator — National Institute of Cardiology; Rafal Dabrowski, MD, PhD, Principal Investigator — National Institute of Cardiology
Locations (1):
- National Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided